CLINICAL TRIAL: NCT00716716
Title: A Phase I/IIa Safety and Pharmacokinetic Study of Intravenous FIXFc in Previously Treated Hemophilia B Patients
Brief Title: Phase I/IIa Study of FIXFc in Hemophilia B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Collaborators: Syntonix Pharmaceuticals, Inc. (Industry); Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYN-FIXFc-07-001
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-08

CONDITIONS: Hemophilia B
Keywords: Hemophilia B severe, previously treated patients
MeSH Terms: conditions — Hemophilia B | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rFIXFc (Experimental): Six intravenous (IV) dose levels, 1, 5, 12.5, 25, 50, and 100 IU/kg
  Interventions: Drug: rFIXFc

INTERVENTIONS:
Drug: rFIXFc — As specified in the treatment arm
  Other Names: Alprolix; recombinant factor IX fusion protein; BIIB029; FIXFc

SUMMARY:
The primary objective of the study is to assess safety of FIXFc at doses ranging from 1 to 100 IU/kg.

DETAILED DESCRIPTION:
This study was previously posted by Syntonix Pharmaceuticals, Inc. In January, 2007, sponsorship of the trial was transferred to Biogen Idec. In February, 2017, sponsorship of the trial was transferred to Bioverativ.

ELIGIBILITY:
Key Inclusion Criteria:

1. Are previously treated (PTPs) with severe (<2 IU/dL endogenous FIX level) hemophilia B and at least 150 prior documented exposure days to other FIX products.
2. Have no prior history of or currently detectable inhibitor defined as > 0.6 Bethesda units by the local lab. A family history of inhibitors will not exclude the patient.
3. No prior history of an allergic reaction or anaphylaxis associated with any FIX or IVIG administration.
4. No concurrent autoimmune disease.
5. At least 7 days since their last dose of FIX (wash-out period).
6. Certain laboratory testing criteria and other protocol-defined criteria may apply.
7. HIV negative or if HIV positive with a CD4 count ≥ 200 cells/mm3. HIV patients are allowed to receive protease inhibitors per the discretion of the Investigator.

Key Exclusion Criteria:

1. Presence of a major bleeding episode on Day 1 of study.
2. Any coagulation disorder in addition to hemophilia B.
3. A patient currently on a dose and regimen of FIX that would preclude participation in the study due to possible increased risk of bleeding because of the requirement to withhold treatment during the study period.
4. A positive d-dimer at screening.
5. Documented history of liver cirrhosis.
6. Positive for HBsAg and/or positive for hepatitis C antibody, and/or HIV positive with an ALT or AST greater than 5 times upper limit of normal.
7. Certain prior illnesses and other protocol-defined criteria.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing Adverse Events | Up to 45 days

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) | Up to 45 days
Maximum concentration (Cmax) | Up to 45 days
Half-life (t½) | Up to 45 days
Clearance (CL) | Up to 45 days
Volume of distribution (Vd) | Up to 45 days
Area under the curve (AUC) | Up to 45 days
Mean residence time (MRT) | Up to 45 days
Incremental recovery (K) | Up to 45 days
Factor IX protein (FIX) activity | Up to 45 days
Recombinant (FIXFc) concentration over time curves | up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (6):
- United States (6):
  - RUSH University Medical Center, Chicago, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of North Carolina Medical School, Chapel Hill, North Carolina
  - Hemophilia Center of Western PA, Pittsburgh, Pennsylvania
  - Puget Sound Blood Center, Seattle, Washington

REFERENCES:
- [Derived] Shapiro AD, Ragni MV, Valentino LA, Key NS, Josephson NC, Powell JS, Cheng G, Thompson AR, Goyal J, Tubridy KL, Peters RT, Dumont JA, Euwart D, Li L, Hallen B, Gozzi P, Bitonti AJ, Jiang H, Luk A, Pierce GF. Recombinant factor IX-Fc fusion protein (rFIXFc) demonstrates safety and prolonged activity in a phase 1/2a study in hemophilia B patients. Blood. 2012 Jan 19;119(3):666-72. doi: 10.1182/blood-2011-07-367003. Epub 2011 Nov 22. PMID 22110246